CLINICAL TRIAL: NCT06041516
Title: A First-in-Human Phase I Trial With Antibody Drug Conjugate ADCT-701 in Neuroendocrine Tumors and Carcinomas
Brief Title: Antibody Drug Conjugate ADCT-701 in Neuroendocrine Tumors and Carcinomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001547; 001547-C
Record Dates: First submitted 2023-09-15; First posted 2023-09-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07-09

CONDITIONS: Neuroendocrine Carcinomas; Neuroendocrine Tumors; Carcinoma, Neuroendocrine; Carcinoma, Adrenocortical; Carcinoma, Adrenal Cortical
Keywords: Pheochromocytoma; Neuroblastoma; Neuroendocrine Tumor; Neuroendocrine carcinoma; Neuroendocrine neoplasms; Paraganglioma; Adrenocortical Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Neuroendocrine Tumors; Adrenocortical Carcinoma; Pheochromocytoma; Neuroblastoma; Paraganglioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Arm1 (Experimental): ADCT-701 given as an IV infusion
  Interventions: Drug: ADCT-701

INTERVENTIONS:
Drug: ADCT-701 — ADCT-701 in 2microgram/kg-255microgram/kg (weight based dosing), IV over 30 minutes (+15 minutes)

SUMMARY:
Background:

Neuroendocrine neoplasms (NENs) are rare cancers in the gastrointestinal tract, pancreas, lungs, adrenal glands, and other areas of the body. Many of these cancers have a high risk of relapse and a low chance of survival. Better treatments are needed.

Objective:

To test a new drug, ADCT-701, in people with NENs.

Eligibility:

Adults aged 18 and older with NENs.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests. They will have imaging scans and tests of heart functioning. Their ability to perform normal daily activities will be tested. A biopsy may be needed: A sample of tissue will be removed from the tumor.

ADCT-701 is given through a tube attached to a needle inserted into a vein in the arm. Participants will receive the drug treatment on the first day of 21-day treatment cycles. They will visit the clinic a total of 10 times during the first two cycles. After that, they will visit the clinic 2 times during each cycle. Imaging scans, blood draws, heart function tests, and other tests will be repeated during study visits. Each visit will last up to 8 hours.

Participants may continue receiving treatment with the study drug for up to 2 years.

After treatment ends, participants will have follow-up clinic visits 4 times in 4 months. They will have a physical exam, with heart and blood tests, at each visit. After that, they will have follow-up clinic visits every 9 weeks; these visits will include imaging scans.

Follow-up visits will continue for up to 5 years after treatment began....

DETAILED DESCRIPTION:
Background:

-Neuroendocrine neoplasms (NENs) are divided into neuroendocrine tumors (NETs) and neuroendocrine carcinomas (NECs). These are rare malignancies occurring in areas such as the gastrointestinal tract, islets of the pancreas, lung, adrenal gland, and other areas of

the body.

* Poorly differentiated neuroendocrine carcinomas are all high-grade carcinomas that resemble small-cell lung cancer (SCLC). Poorly differentiated NECs are also treated with platinum-based regimens in accordance with small cell carcinoma guidelines and have a high risk of relapse as well as a poor response to further systemic therapies.
* Adrenocortical carcinoma (ACC) is a rare malignancy with an average survival from the time of diagnosis of 14.5 months. In advanced diseases, chemotherapy options have limited benefits. To date, no "targeted therapy" has been shown to have significant efficacy in this disease.
* Pre-clinical studies have shown that Delta-like non-canonical notch ligand 1 (DLK1) is expressed in multiple neuroendocrine neoplasms such as ACC, SCLC, neuroblastoma, pheochromocytoma, and paraganglioma.
* ADCT-701 a humanized antibody directed against DLK1 effectively suppresses tumor growth and improves survival in multiple cancer models which express DLK1.

Objective:

-To determine the maximum tolerated dose (MTD) of ADCT-701 in participants with neuroendocrine neoplasms or malignant adrenocortical carcinoma

Eligibility:

* Histologically or cytologically confirmed neuroendocrine neoplasms or malignant ACC.
* Age >= 18 years.
* Evaluable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Adequate organ and bone marrow function.
* Eastern Cooperative Oncology Group (ECOG) <= 2.

Design:

* This is a First in Human phase I dose escalation study of ADCT-701-single agent in participants with NENs.
* Participants will be enrolled in a dose-finding trial. A 3+3 design with up to ten dose levels of ADCT-701 will be evaluated in this trial. The study drug dose will be escalated unless the occurrence of dose-limiting toxicities limits further escalation or until the maximum tolerated dose level is reached or an optimal dose is determined.
* Up to 70 evaluable patients will be enrolled over a maximum of 10 dose levels.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed neuroendocrine neoplasms or malignant adrenocortical carcinoma (ACC).
* Locally advanced or metastatic disease (as confirmed by a radiological evaluation).
* Participants must have measurable disease per RECIST 1.1.
* Participants must have received prior standard of care treatment and be refractory to or intolerant to standard of care therapy(s).
* Age >= 18 years.
* ECOG performance status <= 2.
* Adequate hematologic function as follows:

  * Leukocytes >= 3,000/microliter
  * Absolute neutrophil count (ANC) >= 1,200/microliter (off-growth factors for 72 hours prior to treatment initiation)
  * Hemoglobin (Hgb) >= 9 g/dL with no blood transfusion within 2 weeks prior to treatment initiation
  * Platelets >= 100,000/microliter with no platelet transfusion within 1 week.
* Adequate renal and hepatic function as follows:

  * Creatinine clearance (CrCl) >= 50 mL/min/1.73 m^2 (calculated CrCl (Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) or calculated eGFR provided by a laboratory))
  * Total bilirubin <= 1.5 x ULN OR in participants with known or suspected Gilbert's syndrome, total bilirubin <= 3.0 x ULN
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 2.5 x ULN, (unless liver metastases are present, then values must be <= 5 x ULN).
* Participants serologically positive for hepatitis C virus (HCV) must have an undetectable HCV viral load.
* Participants serologically positive for Hepatitis B (HBV) core antibody or surface antigen must be on adequate anti-viral therapy and Hepatitis B Viral deoxyribonucleic acid (DNA) load must be <2000 IU/mL.
* Participants serologically positive for human immunodeficiency virus (HIV) must be on stable antiretroviral therapy for at least 4 weeks before treatment initiation, have no reported opportunistic infections or Castleman s disease within 12 months prior to treatment initiation, have a viral load that is undetectable by quantitative polymerase chain reaction (PCR) and CD4 count >= 200 cells per cubic millimeter.
* Participants with brain metastasis are eligible if at least 4 weeks status post radiotherapy or surgery before treatment initiation with no evidence of progression or associated symptoms.
* Individuals of child-bearing potential (IOCBP) must agree to use a highly effective method of contraception (hormonal, intrauterine device (IUD), surgical sterilization) for the duration of the study treatment and up to 9.5 months after the last dose of the ADCT-701 (restriction period).

Individuals who can father children must agree to use an effective method of contraception (barrier, surgical sterilization) at study entry and up to 6.5 months after the last dose of the ADCT-701.

* Nursing participants must be willing to discontinue nursing from study treatment initiation through 6.5 months after study treatment discontinuation.
* Participants must be able to understand and be willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Major surgery, prior treatment with chemotherapy, hormonal therapy, immunotherapy, treatment with an investigational agent, and/or radiation therapy within 4 weeks or 5 halflives, whichever is shorter, prior to treatment initiation.
* Participants taking any herbal supplements within 14 days prior to treatment initiation.
* Participants who have wound dehiscence from prior surgeries.
* Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or any serosal effusion that is either requires drainage or is associated with shortness of breath) at screening.
* Active infection requiring systemic antibiotic therapy at screening.
* Active bleeding diathesis or therapeutic anticoagulation with an oral vitamin K antagonist with target international normalized ratio (INR) > 2 at screening.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drug.
* An active autoimmune disease. Note: Participants with type 1 diabetes, eczema, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease, adrenal insufficiency on systemic oral corticosteroid therapy (<= the equivalent of prednisone 10 mg/day), or other mild autoimmune disorders (Type 1 diabetes, eczema, vitiligo, alopecia, rheumatoid arthritis, psoriasis, systemic lupus erythematosus, adrenal insufficiency due to Addison s disease, hypothyroidisms due to Hashimoto s thyroiditis, hyperthyroidisms due to Graves disease, Sjogren s syndrome, celiac disease, pernicious anemia) not requiring immunosuppressive treatment are eligible.
* Congenital long QT syndrome, or a corrected QTcF interval of >=480 ms, at screening (unless secondary to the pacemaker or bundle branch block).
* Active second primary malignancy other than non-melanoma skin cancers, nonmetastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that does not require current anticancer treatment per standard of care.
* Live vaccine administration within 30 days prior to treatment initiation.
* Pregnant individuals (confirmed by Beta-Human Chorionic Gonadotropin [Beta-HCG] serum or urine pregnancy test) performed at screening.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of ADCT-701 | cycle 1, days 1-21
  Number of dose-limiting toxicities (DLTs) by assessing adverse events (AE) by type and grade of toxicity.

SECONDARY OUTCOMES:
Safety of ADCT-701 | through 30 days after the last ADCT-701 infusion
  Adverse Events (AE) by type and grade of toxicity
Preliminary anti-tumor activity of ADCT-701 | up to 5 years
  To capture response rate and durations to assess: overall response rate (ORR), duration of response (DOR), progression-free survival (PFS), and overall survival (OS)
PK profile of ADCT-701 | up to 2 years
  Assessment of PBD-conjugated antibody, total antibody, and unconjugated warhead SG3199 in blood.
Immunogenicity of ADCT-701 | up to 2 years
  Assessment of ADAs using a screening assay for the identification of antibody-positive samples, a confirmation assay, and a titer assessment in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Jaydira Del Rivero, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI

REFERENCES:
- [Derived] Sun NY, Kumar S, Kim YS, Varghese D, Mendoza A, Nguyen R, Okada R, Reilly K, Widemann B, Pommier Y, Elloumi F, Dhall A, Taniyama D, Patel M, Aber E, Contreras CF, Kaplan RN, Kiseljak-Vassiliades K, Wierman ME, Martinez D, Pogoriler J, Hamilton AK, Diskin SJ, Maris JM, Robey RW, Gottesman MM, Del Rivero J, Roper N. Identification of the Notch ligand DLK1 as an immunotherapeutic target and regulator of tumor cell plasticity and chemoresistance in adrenocortical carcinoma. Nat Commun. 2025 Jul 1;16(1):5511. doi: 10.1038/s41467-025-60649-w. PMID 40595495
- [Derived] Sun NY, Kumar S, Kim YS, Varghese D, Mendoza A, Nguyen R, Okada R, Reilly K, Widemann B, Pommier Y, Elloumi F, Dhall A, Patel M, Aber E, Contreras-Burrola C, Kaplan R, Martinez D, Pogoriler J, Hamilton AK, Diskin SJ, Maris JM, Robey RW, Gottesman MM, Rivero JD, Roper N. Identification of DLK1, a Notch ligand, as an immunotherapeutic target and regulator of tumor cell plasticity and chemoresistance in adrenocortical carcinoma. bioRxiv [Preprint]. 2024 Oct 11:2024.10.09.617077. doi: 10.1101/2024.10.09.617077. PMID 39416174
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001547-C.html